CLINICAL TRIAL: NCT00897819
Title: Evaluation of the Association Between DNA Methylation and Shortened Survival in Patients With Advanced Colorectal Cancer Treated With 5-FU/Oxaliplatin-Based Regimens in E3200
Brief Title: Studying DNA and Outcome in Patients With Advanced Colorectal Cancer Treated With Fluorouracil and Oxaliplatin With or Without Bevacizumab on Clinial Trial E-3200
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000534281; ECOG-E3200T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer; stage III colon cancer; stage III rectal cancer; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: loss of heterozygosity analysis
Genetic: microsatellite instability analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood, urine, and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This laboratory study is analyzing the DNA in tissue samples from patients with advanced colorectal cancer treated with fluorouracil and oxaliplatin with or without bevacizumab on clinical trial E-3200.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the CpG island methylation pathway markers that are adverse for survival after treatment with fluorouracil in patients with advanced colorectal adenocarcinoma treated with fluorouracil and oxaliplatin with or without bevacizumab on clinical trial E-3200.
* Compare the methylation results to clinicopathologic and molecular findings and survival.

OUTLINE: This is a multicenter study.

Tissue, blood, and urine samples and genomic DNA samples from tumor tissue blocks are examined by pyrosequencing assay for methylation. Genes examined include MINT1, MINT31, P14, and P16. Microsatellite instability and loss of heterozygosity (LOH) on chromosome 18 (18q LOH) are also assessed. Microsatellites examined include BAT loci, TGFβRII, D2S123, D55346, and D17S250.

PROJECTED ACCRUAL: A total of 350 specimens will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the colon or rectum

  * Advanced disease
* Enrolled on clinical trial E-3200 and received fluorouracil and oxaliplatin
* Tumor tissue blocks available
* Routine pathology specimens (i.e., blood, urine) available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E3200
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2007-01-03 (Actual); Primary Completion 2008-01-30 (Actual); Study Completion 2008-01-30 (Actual)

PRIMARY OUTCOMES:
Correlation of MSI and LOH to outcome and response | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hamilton, MD, Study Chair — M.D. Anderson Cancer Center